CLINICAL TRIAL: NCT01861977
Title: Healthy Habits Program for High Cardiovascular Risk Patients: Randomized Controlled Clinical Trial. Effectiveness of a Program Using Cognitive Behavioral Therapy to Improve Healthy Habits in a Population With Cardiovascular Disease.
Brief Title: Healthy Habits Program for High Cardiovascular Risk Patients: Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Gaston Perman, Head of Medical Programs, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009
Record Dates: First submitted 2013-05-21; First posted 2013-05-24 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior; Motor Activity; Food Habits
Keywords: Cognitive Therapy; Health Education; Secondary Prevention; Cardiovascular Disease
MeSH Terms: conditions — Health Behavior; Motor Activity; Feeding Behavior; Health Education; Cardiovascular Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Participants in this arm will be invited to attend 8 weekly group meetings and 3 monthly follow-up meetings. In each meeting a coordinator will explore the experiences of the participants and encourage them to look for strategies to solve problems associated with changing habits. In the meetings we will use a therapeutic education approach with motivational interviewing techniques and problem solving in order to increase self-efficacy and motivation to adopt healthy habits. There will be periodic reminders and telephone contacts with patients before the meetings to assess the achievement of objectives.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Informational Workshop (Active Comparator): Participants will be invited to participate in 4 weekly group meetings and an additional reinforcing meeting in the 5th month. In each meeting, workshop techniques will be used, together with educational materials as brochures, pictures, etc. The informational material will focus on the benefits of lifestyle changes in diet and physical activity.
  Interventions: Behavioral: Informational Workshop

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants in this arm will be invited to attend 8 weekly group meetings and 3 monthly follow-up meetings. In each meeting a coordinator will explore the experiences of the participants and encourage them to look for strategies to solve problems associated with changing habits. In the meetings we will use a therapeutic education approach with motivational interviewing techniques and problem solving in order to increase self-efficacy and motivation to adopt healthy habits. There will be periodic reminders and telephone contacts with patients before the meetings to assess the achievement of objectives.
  Arms: Cognitive Behavioral Therapy
Behavioral: Informational Workshop — Participants will be invited to participate in 4 weekly group meetings and an additional reinforcing meeting in the 5th month. In each meeting, workshop techniques will be used, together with educational materials as brochures, pictures, etc. The informational material will focus on the benefits of lifestyle changes in diet and physical activity.
  Arms: Informational Workshop

SUMMARY:
The purpose of this study is to determine the effectiveness of a program to improve habits in a population with cardiovascular disease, comparing two different educational techniques (cognitive behavioral therapy group vs. informational workshops).

ELIGIBILITY:
Inclusion Criteria:

* Patients who live in the catchment area of the health centers participating in the trial or that have their primary care physician in these centers.

or

* Patients with a diagnosis of coronary heart disease, and / or transluminal angioplasty and / or coronary artery bypass grafting (CABG). These diagnoses must have occurred longer than six months from the time of inclusion.

or

* Patients with a diagnosis of cerebrovascular accident (CVA), transient ischemic attack (TIA), carotid endarterectomy and / or carotid angioplasty. These diagnoses must have occurred longer than six months from the time of inclusion.

or

* Patients with peripheral arterial disease with or without intermittent claudication, revascularization surgery, bypass placement of arterial and / or peripheral arterial angioplasty. These diagnoses must have occurred longer than six months from the time of inclusion.

and

* Sedentary persons, defined as less than 90 minutes per week of moderate aerobic physical activity in their daily life (leisure, travel or work).

Exclusion Criteria:

- Patients on chronic home monitoring and / or institutionalized before admission or living in a tertiary institution.

or

* Moderate or severe limitation on functional capacity and / or mobility. or
* Patients with dementia. or
* Patients diagnosed with psychiatric illnesses that compromise patient autonomy. or
* Life expectancy less than 1 year. or
* Patients who do not want to take part in the program. or
* Patients who are participating in another research protocol at recruitment. or
* Patients with a diagnosis of intracranial hemorrhage secondary to aneurysmal rupture.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Achievement of moderate physical activity recommendations | One year
  Moderate physical activity: minutes per week measured by the questionnaire WHO STEP wise (Physical activity at work/in the household, for transport and during leisure time; minimum 0; the grater the better).
Consumption of fruits and vegetables | One year
  Consumption of fruits and vegetables: number of servings per day measured by questionnaire WHO STEP wise (minimum 0; optimal 5 or more).

SECONDARY OUTCOMES:
Smoking cessation | One year
  Smoking cessation: will be considered if patients report smoking abstinence (no smoking consumption for the last three months), at the end of the study.
Blood pressure control | One year
  Blood pressure will be considered controlled if systolic blood pressure values are lower than 140 mmHg and/or if there is a decrease in at least 5% from basal at the end of the program.
Lipid Control | One year
  LDL cholesterol will be considered controlled if the patient has LDL values below 100 mg/dl or a reduction of at least 20% from basal at the end of the program.
Body weight reduction | One year
  Reducing at least 5% from basal of body weight at endpoint in those patients with a body mass index (BMI) in a value greater than 30 kg/m2 at baseline.

OTHER OUTCOMES:
Improvement in health related quality of Life | One year.
  Perception of quality of life will be assessed through EuroQol questionnaire (validated in Spanish). It will analyze the difference (final-basal) between the two groups. The visual analog scale ranges from 0 (worse quality of life possible) to 100 (best possible state).
Treatment Adherence | One year
  Maintaining adherence to prescribed drug treatments: adherence to drug treatment will be evaluated through Medication Adherence Questionnaire. It will analyze the final difference (final-basal) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gaston Perman, MD, MSc, Study Director — Hospital Italiano de Buenos Aires; Gabriela Buela, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186
- [Background] Lim HK, Foltz RL. In vivo formation of aromatic hydroxylated metabolites of 3,4-(methylenedioxy)methamphetamine in the rat: identification by ion trap tandem mass spectrometric (MS/MS and MS/MS/MS) techniques. Biol Mass Spectrom. 1991 Nov;20(11):677-86. doi: 10.1002/bms.1200201105. PMID 1686830
- [Background] Ismail K, Winkley K, Rabe-Hesketh S. Systematic review and meta-analysis of randomised controlled trials of psychological interventions to improve glycaemic control in patients with type 2 diabetes. Lancet. 2004 May 15;363(9421):1589-97. doi: 10.1016/S0140-6736(04)16202-8. PMID 15145632
- [Background] Berkman LF, Blumenthal J, Burg M, Carney RM, Catellier D, Cowan MJ, Czajkowski SM, DeBusk R, Hosking J, Jaffe A, Kaufmann PG, Mitchell P, Norman J, Powell LH, Raczynski JM, Schneiderman N; Enhancing Recovery in Coronary Heart Disease Patients Investigators (ENRICHD). Effects of treating depression and low perceived social support on clinical events after myocardial infarction: the Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Randomized Trial. JAMA. 2003 Jun 18;289(23):3106-16. doi: 10.1001/jama.289.23.3106. PMID 12813116
- [Background] Gulliksson M, Burell G, Vessby B, Lundin L, Toss H, Svardsudd K. Randomized controlled trial of cognitive behavioral therapy vs standard treatment to prevent recurrent cardiovascular events in patients with coronary heart disease: Secondary Prevention in Uppsala Primary Health Care project (SUPRIM). Arch Intern Med. 2011 Jan 24;171(2):134-40. doi: 10.1001/archinternmed.2010.510. PMID 21263103
- [Background] Smith SC Jr, Benjamin EJ, Bonow RO, Braun LT, Creager MA, Franklin BA, Gibbons RJ, Grundy SM, Hiratzka LF, Jones DW, Lloyd-Jones DM, Minissian M, Mosca L, Peterson ED, Sacco RL, Spertus J, Stein JH, Taubert KA. AHA/ACCF secondary prevention and risk reduction therapy for patients with coronary and other atherosclerotic vascular disease: 2011 update: a guideline from the American Heart Association and American College of Cardiology Foundation endorsed by the World Heart Federation and the Preventive Cardiovascular Nurses Association. J Am Coll Cardiol. 2011 Nov 29;58(23):2432-46. doi: 10.1016/j.jacc.2011.10.824. Epub 2011 Nov 3. No abstract available. PMID 22055990
- [Background] Furie KL, Kasner SE, Adams RJ, Albers GW, Bush RL, Fagan SC, Halperin JL, Johnston SC, Katzan I, Kernan WN, Mitchell PH, Ovbiagele B, Palesch YY, Sacco RL, Schwamm LH, Wassertheil-Smoller S, Turan TN, Wentworth D; American Heart Association Stroke Council, Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the prevention of stroke in patients with stroke or transient ischemic attack: a guideline for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Jan;42(1):227-76. doi: 10.1161/STR.0b013e3181f7d043. Epub 2010 Oct 21. PMID 20966421
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Result] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Result] Barth J, Schneider S, von Kanel R. Lack of social support in the etiology and the prognosis of coronary heart disease: a systematic review and meta-analysis. Psychosom Med. 2010 Apr;72(3):229-38. doi: 10.1097/PSY.0b013e3181d01611. Epub 2010 Mar 11. PMID 20223926
- [Result] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889